CLINICAL TRIAL: NCT06732635
Title: Enhanced Recovery After Surgery (ERAS) for Laparoscopic Hysterectomy at Low Risk Endometrial Cancer: A Randomized Controlled Trial
Brief Title: Enhanced Recovery After Surgery (ERAS) for Laparoscopic Hysterectomy at Low Risk Endometrial Cancer
Acronym: FAST-TRACK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAS
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: A controlled, randomized, parallel-group, open-label, interventional, single-center clinical trial in which the intervention group will be managed according to the multimodal rehabilitation protocol (RICA clinical pathway), and the control group will receive traditional care that has been provided up to now.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention)
- ERAS (Experimental): Enhanced recovery after surgery (ERAS) programs are designed to achieve early recovery after surgery and a shorter length of stay (LOS) at hospital.
  Interventions: Procedure: Enhanced recovery after surgery (ERAS)

INTERVENTIONS:
Procedure: Enhanced recovery after surgery (ERAS) — Enhanced recovery after surgery (ERAS) programs are designed to achieve early recovery after surgery and a shorter length of stay (LOS) at hospital.
  Arms: ERAS

SUMMARY:
Enhanced recovery after surgery (ERAS) programs are designed to achieve early recovery after surgery and a shorter length of stay (LOS) at hospital.

So far there are only three prospective, randomised studies that exclusively analyze patients affected by oncogynecological pathology providing a high level of scientific evidence. To our knowledge, no studies have been conducted specifically on ERAS pathways in endometrial cancer treated by laparoscopy. This study aims to evaluate whether ERAS pathways are beneficial for patients with endometrial cancer, particularly among low-risk early endometrial cancer operated by laparoscopy. Length of stay (LOS), perioperative morbidity and mortality, and perioperative quality of life were analyzed comparing both ERAS and Conventional protocols groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic hysterectomy for stage 1A and 1B endometrial cancer

Exclusion Criteria:

* Age under 18 years
* ASA IV
* Liver cirrhosis
* Psychiatric illness
* Urgent surgery
* The patient's desire not to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Lengh of stay | 30 days after surgery
  Days of hospitalitation
Day of discharge | 30 days after surgery
Readmisión | During 1st month after surgery
  yes/no

OTHER OUTCOMES:
Complications | 30 days after surgery
  Clavien-Dindo Classification. Scale rated from grade 1 to grade 5 The Clavien-Dindo (CD) classification is widely used in the reporting of surgical complications in scientific literature. It groups complications based on the level of intervention required to resolve them, and benefits from simplicity and ease of use, both of which contribute its to high inter-rater reliability
Quality of life (QoL) | Preoperative, 3, 10 and 30 days after surgery
  Core Quality of Life questionnaire (EORTC QLG Core Questionnaire) (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients. You should select the option that best represents you from the options 1Not at All, 2A little, 3Quite a bit, 4Very much
Level of Pain | Preoperative, 3, 10 and 30 days after surgery
  Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain